CLINICAL TRIAL: NCT01879293
Title: Metformin Reduces Left Ventricular Mass in Patients With Ischemic Heart Disease:A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Metformin Reduces Left Ventricular Mass in Patients With Ischemic Heart Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wuhan General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Xiang Guang-da, Director of Endocrinol Dept., Wuhan General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2013Wze028
Record Dates: First submitted 2013-06-11; First posted 2013-06-17 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Left Ventriclar Mass
Keywords: Metformin; Left ventricular mass; Endothelial dysfunction; cardiac magnetic resonance; aortic pulse wave
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin group (Experimental): In this group, metformin 0.5 three times daily for one year.
  Interventions: Drug: Metformin
- Placebo group (Placebo Comparator): In this group, placebo will be given twice daily for one year.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Metformin
  Arms: Metformin group
Drug: placebo
  Arms: Placebo group

SUMMARY:
Cardiovascular disease is the most common cause of death in the world. Most of the attention in treating ischemic heart disease (IHD) is understandably directed toward treating coronary artery disease. However there are other treatable culprits in these patients.

Left ventricular hypertrophy (LVH) is widespread in IHD patients, even in the absence of hypertension. It is a strong predictor of cardiovascular events and all-cause mortality. In one study, the presence of LVH was a stronger predictor of mortality than either multivessel cor-onary disease or impaired LV function.

Metformin is an antihyperglycemic agent with a history of successful use in type 2 diabetes. In the UKPDS (United Kingdom Prospective Diabetes Study), metformin was associated with a 39% lower risk of myocardial infarction compared with conventional therapy. Metformin also offered dual benefits of improving vascular function and lessening ischemia in nondiabetic patients.

Hence, the main aim of this study was to assess whether metformin could regress LVM in patients with IHD. The secondary aim was to assess the effect of metformin on LV volumes and endothelial function in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* They had to have normal glucose tolerance.
* They had to have either angiographically documented coronary artery disease or a previous history of myocardial infarction.
* They were required to have an office BP < 130/80 mm Hg
* The presence of LVH on echocardiography (American Society of Echocardiography criteria LVM index [LVMI] > 115 g/m2 for men and > 95 g/m2 for women).

Exclusion Criteria:

* They were currently prescribed metformin.
* They had renal and liver dysfunction, heart failure, or malignancy, or were unable to give informed consent.
* Patients with contraindications to cardiac magnetic resonance (CMR) (pacemakers, claustrophobia) were also excluded, as were pregnant or lactating women.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Left ventricular mass. | one year
  We will measure left ventricular mass before and after metformin intervention with cardiac magnetic resonance.

SECONDARY OUTCOMES:
Left ventricular volume and endothelial function. | one year
  We measure the left ventricular volume and endothelial function before and after metformin intervention by cardiac magnetic resonance and high resolution ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan General Hospital, Wuhan, Hubei, China